CLINICAL TRIAL: NCT06371287
Title: Effect of Musical Auditory Training on Neuroplasticity and Perception of Subjects With Tinnitus Disorder
Brief Title: Effect of Musical Auditory Training on Subjects With Tinnitus Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Christine Grellmann Schumacher, Investigator Official, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 64696022.1.0000.5346
Record Dates: First submitted 2024-02-27; First posted 2024-04-17 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Tinnitus
Keywords: Plasticidade Neuronal; Zumbido; Processamento Auditivo Central
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group - Musical Auditory Training (Experimental): For musical training, the protocol proposed by Freire, et al. (2009). This protocol was created for elderly users of hearing aids and in this study it will be used as an instrument for intervention in tinnitus, aiming at auditory training through the hierarchization of auditory skills associated with musicality (FREIRE, 2009).
  Eight sessions will be held over four weeks, two sessions per week. Sessions will last a minimum of 40 minutes and a maximum of 50 minutes. Victory supra-aural headphones will be used, connected to the computer. There will be calibration, with adjustment of the volume of sounds to the most comfortable level for the individual at the beginning of all sessions.
  Interventions: Behavioral: Treinamento Auditivo Musical
- Control Group - Placebo (Placebo Comparator): Placebo sessions will also be held twice a week for four weeks, totaling eight sessions.
  To ensure the same conditions for performing musical auditory training, in the placebo treatment, instrumental music will be used concomitantly with the exposure of films without sound, in which patients will be exposed to visual and auditory stimulation during the same time of EG intervention, at least 40 minutes and a maximum of 50 minutes.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Treinamento Auditivo Musical — Auditory training with a focus on musicality. The skills trained will be: figure-ground for instrumental sounds, sequential figure-ground, directed listening, duration of sounds, frequency of sounds, rhythm (temporal structuring), auditory closure and audiovisual memory, with a focus on temporal processing, working memory and attention selective on an increasing scale of difficulty. The frequency ranges of instrumental sounds are from 200 to 4000 Hz, composed of the following instruments: guitar, vibraphone, piano, flute and drum.
  Arms: Study Group - Musical Auditory Training
Behavioral: Placebo — This placebo approach will be to demonstrate the influence of musical exposure without exercises with structuring auditory skills and compare with the TAM group.
  The song Sonata for two pianos in D major, K448, by Mozart, will be used. The films selected were: Cirque Du Soleil, entitled "The Journey of Man"; Chaplin collection with the following films: "Modern Times", "The Great Dictator", "In Search of Gold" and "Footlights". The choice of the order of the films will be random, as proposed by Freire (2009).
  Arms: Control Group - Placebo

SUMMARY:
Among the theories of tinnitus generation, there is that of central neuroplastic changes, which reports the association between changes and reorganization that occur in central auditory pathways and impacts on associated areas due to the altered neural signal. Auditory training modifies these altered pathways through auditory exercises, which provoke positive neuroplasticity. Musical auditory training is a proposal to stimulate auditory, cognitive and metalinguistic skills with activities focused on musicality. Therefore, the objective of this study is to verify the effect of musical auditory training (MAT) on the neuroplasticity of the auditory system and the perception of tinnitus disorder in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes aged between 18 years and 55 years;
* Complaint of chronic tinnitus (minimum perception of six months) unilateral or bilateral;
* Hearing thresholds within normal limits bilaterally or even mild sensorineural hearing loss in the four-tone average (500, 1000, 2000 and 4000Hz);
* Annoyance score of at least four on the Visual Analogue Scale, considered a moderate symptom discomfort;
* Have normality in the Mini Mental State Examination (cognitive screening).

Exclusion Criteria:

* Apparent speech, psychiatric or neurological changes;
* History of head or brain trauma;
* Objective tinnitus (somatosensory and vascular);
* Present symptoms and/or diagnosis of middle ear involvement;
* Having started a new treatment (pharmacological or therapeutic) or having been diagnosed with a disease of any origin in the last month.
* Be carrying out another intervention for tinnitus during the research;
* Use of electronic assistive hearing devices.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Changes in latency of the long latency auditory evoked potential (LLAEP) | Within a month
  Improve the latency in milliseconds of P2 potential

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No